CLINICAL TRIAL: NCT01520831
Title: A Randomised, Four-period Cross-over Trial in Healthy Subjects, Investigating the Pharmacodynamics and Pharmacokinetics of Biphasic Insulin Aspart 30, Biphasic Insulin Aspart 50, Biphasic Insulin Aspart 70 and Soluble Insulin Aspart
Brief Title: Comparison of Biphasic Insulin Aspart (30, 50 and 70) and Insulin Aspart in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BIASP-1086
Record Dates: First submitted 2012-01-25; First posted 2012-01-30 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- BIAsp 30 (Experimental)
  Interventions: Drug: biphasic insulin aspart 30
- BIAsp 50 (Experimental)
  Interventions: Drug: biphasic insulin aspart 50
- BIAsp 70 (Experimental)
  Interventions: Drug: biphasic insulin aspart 70
- Insulin aspart (Active Comparator)
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — One single dose of 0.3 U/kg body weight administered subcutaneously (s.c., under the skin) at one of four study days
  Arms: BIAsp 30
Drug: biphasic insulin aspart 50 — One single dose of 0.3 U/kg body weight administered subcutaneously (s.c., under the skin) at one of four study days
  Arms: BIAsp 50
Drug: biphasic insulin aspart 70 — One single dose of 0.3 U/kg body weight administered subcutaneously (s.c., under the skin) at one of four study days
  Arms: BIAsp 70
Drug: insulin aspart — One single dose of 0.3 U/kg body weight administered subcutaneously (s.c., under the skin) at one of four study days
  Arms: Insulin aspart

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to demonstrate a difference between the pharmacodynamics and pharmacokinetics of biphasic insulin aspart 30, biphasic insulin aspart 50, biphasic insulin aspart 70 and insulin aspart in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18 and 28 kg/m^2 inclusive
* HbA1c within the normal laboratory range
* Non smoker for at least three months
* Females of childbearing potential using acceptable methods of contraception, including tubal ligation, an intrauterine device (IUD) , the oral contraceptive pill or barrier methods

Exclusion Criteria:

* Subjects who have received any investigational drug in the 3 months prior to the start of dosing
* Any disease requiring regular use of non topical prescription medicines
* Any serious systemic infectious disease that occurred in the 4 weeks prior to the first dose of test drug
* Any intercurrent illness or endocrine disorders that may affect blood glucose
* Subject with a history of drug or alcohol dependence
* Subject with a first degree relative with diabetes mellitus
* Subject with a history of clinically relevant allergic reactions to medical products
* Subjects who have donated any blood or plasma in the past 3 month preceding screening

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 1999-04; Primary Completion 2000-05 (Actual); Study Completion 2000-05 (Actual)

PRIMARY OUTCOMES:
Area under the GIR (Glucose Infusion Rate) profile (AUC GIR) in the interval 0-120 minutes

SECONDARY OUTCOMES:
Maximum GIR value
Time to maximum GIR value
Area under the GIR profile
Cmax, maximum insulin aspart concentration
Area under the insulin aspart concentration curve
tmax, the time to maximum insulin aspart concentration
t½, terminal half-life

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- [Result] Heise T, Kapitza C, Jacobsen LV, Brøndsted L, Heinemann L. Pharmacokinetic and pharmacodynamic differences between premixed suspensions of insulin aspart: biphasic insulin aspart 30, 50 and 70. Diabetologia 2005; 48 (Suppl. 1): A301
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com